CLINICAL TRIAL: NCT02796430
Title: Clinical Evaluation of the Ease of Use of a New Indirect Calorimeter for Energy Expenditure Measurement in ICU Patients: The ICALIC International Multicentric Study
Brief Title: The ICALIC International Multicentric Study
Acronym: ICALIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: European Society of Intensive Care Medicine (Other); European Society for Clinical Nutrition and Metabolism (Other)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Claude Pichard, MD, PhD, University Hospital, Geneva
Other Study IDs: 15-137
Record Dates: First submitted 2016-05-31; First posted 2016-06-10 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Critical Illness
Keywords: Indirect calorimetry; critical care; mechanical ventilation; energy expenditure; ICALIC study
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated patients: Ease of use will be assessed by analysing the time needed to start indirect calorimetry measurement, and results of indirect calorimetry measurements by both the new indirect calorimeter and the currently used calorimeters at each study center.
  Interventions: Other: Time needed to start indirect calorimetry measurement; Other: Indirect calorimetry measurement

INTERVENTIONS:
Other: Time needed to start indirect calorimetry measurement — Comparison of the time needed to start EE measurements by the new calorimeter and the currently used calorimeter, including the time needed for calibration, patient data input, connection to the ventilator circuit.
Other: Indirect calorimetry measurement — Comparison of EE measurements by the new calorimeter and the currently used calorimeter when using different mechanical ventilators, different ventilation modes, different patient conditions and severity

SUMMARY:
This study will evaluate the ease of use of the new calorimeter (Q-NRG (COSMED, Italy)) in intensive care unit (ICU) patients compared to currently used calorimeters (i.e. Quark RMR 1.0(COSMED, Italy) or Deltatrac Metabolic Monitor (Datex, Finland)), as well as the stability and the feasibility of the measurements in various clinically relevant situations.

Time needed to prepare and start indirect calorimetry (IC) measurement will be compared as the measure of the ease of use of the calorimeter.

DETAILED DESCRIPTION:
Background and Aims:

This study aims at evaluating the ease of use of the new calorimeter for the measurement of energy expenditure (EE) in intensive care unit (ICU) patients. EE in ICU patients is highly variable depending on the severity of the disease and treatments. Clinicians need to measure EE by indirect calorimetry (IC) to optimize nutritional support for the better clinical outcome. However, indirect calorimeters available on the market have insufficient accuracy for clinical and research use. Difficulties of handling and interpretation of results often limit IC in ICU patients. An accurate, easy-to-use calorimeter has been developed to meet these needs.

The Study Device:

The new calorimeter (Q-NRG, COSMED) is capable of IC measurements in mechanically ventilated patients without warm-up and limited calibration. The disposable in-line pneumotach flow meter and direct sampling of respiratory gas from the ventilator circuit enables the accurate measurement of oxygen consumption volume (VO2) and CO2 production volume (VCO2) to derive the energy expenditure. The software interface to manage the device and the collected data provides easy-to-use, user-friendly interface. Q-NRG does not bear the European Commission Conformity Mark (CE Mark), but has been approved by the Swiss authority for medical devices (Swissmedic) for use in this study. Q-NRG will be used in the way it is intended to be used as described in the instruction manual.

Currently used indirect calorimeters at each study center will be used as the comparator.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated adult ICU patients

Exclusion Criteria:

* Fraction of inhaled oxygen (FIO2) > 70%
* Positive end expiratory pressure (PEEP) >10cmH2O
* Peak ventilatory pressure > 30cmH2O
* Presence of air leaks from thoracic drain tube
* Changes in vasoactive agent dose (>20%, <1 hr before and/or during IC)
* Agitation or change in sedative dose (>20%, <1 hr before and/or during IC)
* Change in body temperature (>0.5°C, <1 hr before and/or during IC)
* Expected duration of ICU stay < 24 hours
* Expected survival of the patient < 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated adult ICU patients
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Time needed to start indirect calorimetry (IC) measurement in Q-NRG compared to currently used calorimeters | immediately after the measurement
  Time from the start-up of the devices until the 1st recorded measurement will be measured and compared between Q-NRG and the currently used indirect calorimeters, including time needed for patient information input, warm-up and calibrations according to the instructions for the devices, and installation of the device components needed for the measurements on patients.

SECONDARY OUTCOMES:
Comparison of energy expenditure(EE) from Q-NRG and currently used calorimeters | immediately after the measurement
  EE measured by Q-NRG and currently used calorimeters will be compared to identify the differences of the characteristics of the measurements according to the different types of calorimeters.
Coefficient of variation (CV) of EE for different mechanical ventilators | immediately after the measurement
  CV of EE measured by Q-NRG when using different mechanical ventilators will be analyzed to evaluate the effects of the mechanical ventilators used during the indirect calorimetry measurement.
CV of EE when using different ventilation modes | immediately after the measurement
  CV of EE measured by Q-NRG when using different mechanical ventilation modes will be analyzed to evaluate the effect of different mechanical ventilation modes used during the indirect calorimetry measurement.
CV of EE in various ranges of oxygen and airway pressure support | immediately after the measurement
  CV of EE measured by the Q-NRG in different ranges of FiO2 will be analyzed to evaluate the difference in the stability of the measurements according to various FiO2 ranges.
CV of EE when measured in different sedation/consciousness levels | immediately after the measurement
  CV of EE measured by the Q-NRG in different levels of sedation/consciouness will be analyzed to evaluate the difference in the stability of the measurements according to various sedation/consciousness levels.
CV of EE when measured in different levels of patient severity | immediately after the measurement
  CV of EE measured by the Q-NRG in different levels of patient severity will be analyzed to evaluate the difference in the stability of the measurement according to various levels of severity.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichard, MD, PhD, Principal Investigator — Clinical Nutrition, Geneva University Hospital
Locations (7):
- Division of Cardiac Thoracic Vascular Anesthesia and Intensive Care Medicine, Vienna, Austria
- Department of Intensive Care, Vrije Universiteit Brussel, Brussels, Belgium
- Critical Care Medicine, Institute for Nutrition Research, Rabin Medical Center, Beilison Hospital, Petah Tikva, Israel
- Chiba University Hospital, Chiba, Japan
- Department of Anesthesiology and Intensive Care Medicine, Karolinska University Hospital, Huddinge, Sweden
- Switzerland (2):
  - Service of Intensive Care, Geneva University Hospital, Geneva
  - Adult Intensive care, Lausanne University Hospital, Lausanne

IPD SHARING:
Plan to Share IPD: No